CLINICAL TRIAL: NCT05887050
Title: Effects of a Dietary Supplement Containing Salacia Extract, Citrus Bioflavonoids, and Trivalent Chromium on Markers of Glucose Control and Quality of Life: A Randomized, Placebo-Controlled, Double-Blind Pilot Study
Brief Title: Effects of a Dietary Supplement Containing Salacia Extract, Citrus Bioflavonoids, and Trivalent Chromium on Markers of Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MEND-2023
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All participants were randomly assigned to receive either the active product or a placebo. Subjects were instructed to consume their respective supplement daily for 12 weeks, approximately 15-30 minutes prior to their evening meal.
Who Masked: Investigator
Masking Description: Supplements were blinded by the sponsor prior to initiation of any research activities. All research activities, including statistical analysis, were completed by the research team while blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Tablet containing 400 mcg chromium (delivered as Crominex® 3+, a blend of chromium, Capros® Amla Extract (Fruit), PrimaVie® Shilajit), and 325 mg of MetaviveTM complex (Salacia Chinensis Extract (Fruit) and a Citrus Bioflavonoid Complex)
  Interventions: Dietary Supplement: Active
- Placebo (Placebo Comparator): Identical size, shape, and weight maltodextrin tablet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active — Blend of chromium, amla fruit extract, and citrus bioflavonoids
  Arms: Active
Dietary Supplement: Placebo — Maltodextrin tablet
  Arms: Placebo

SUMMARY:
This study was a double-blind, randomized, placebo-controlled, clinical trial with two parallel groups. Participants reported to a single investigational center in Ohio (i.e., The Center for Applied Health Sciences) during the 12 week trial.

DETAILED DESCRIPTION:
This study was a double-blind, randomized, two-arm, placebo-controlled trial of apparently healthy men and women recruited at a single investigational center in Northeast Ohio (i.e. The Center for Applied Health Sciences).

Subjects will attend four study visits. During Visit 1, subjects will be screened for participation (i.e., medical history, physical exam, routine blood work [also HgA1c, insulin], background baseline diet). Over the next 12 weeks, subjects will attend Visits 2-4, wherein assessments of serum glucose, insulin, HOMA-IR, 2-hour glucose tolerance test (GTT), NMR profile, HgA1c, C-reactive protein, adiponectin, ferritin, waist circumference, quality of life questionnaire, and various visual analog scales for appetite, satiety, and cravings will be made (see Study Schematic for details).

Comprehensive side effect profile/ adverse event monitoring will take place throughout the study duration. The study will be conducted following ICH-GCP guidelines to ensure subject safety and scientific integrity of the data.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between the ages of 21 and 65 (inclusive).
* Body Mass Index of 18.5-34.99 (inclusive).
* Body weight of at least 120 pounds.
* Fasting blood sugar of 100-125 (inclusive) OR HgA1c of 5.7-6.4% (inclusive).
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from caffeine for 12 hrs and exercise

Exclusion Criteria:

* History of unstable or new-onset cardiovascular or cardiorespiratory disease.
* History of diabetes, or other endocrine disorder.
* Fasting blood sugar of > 125 mg/dL or HgA1c of > 6.4%.
* History of use of medications or dietary supplements known to affect glycemia or insulinemia.
* History of hyperparathyroidism or an untreated thyroid disease.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband), etc.
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g. short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or disease (e.g. rheumatoid arthritis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of-Analysis.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Glucose kinetics | Change from baseline to 12 weeks.
  Serum glucose response during a two hour oral sucrose tolerance test.
Insulin kinetics | Change from baseline to 12 weeks.
  Serum insulin response during a two hour oral sucrose tolerance test.

SECONDARY OUTCOMES:
Hemoglobin A1c (HgA1c) | Change from baseline to 12 weeks.
  Serum HgA1c
C-reactive protein | Change from baseline to 12 weeks.
  Serum C-reactive protein
Adiponectin | Change from baseline to 12 weeks.
  Serum adiponectin
Ferritin | Change from baseline to 12 weeks.
  Serum ferritin
Appetite | Change from baseline to 12 weeks.
  Appetite as measured by a 10 cm visual analogue scale, where higher values represent greater appetite. Values range from 1-10, and a greater appetite score would be a worse outcome in these participants.
Satiety | Change from baseline to 12 weeks.
  Satiety as measured by a 10 cm visual analogue scale, where higher values represent greater satiety. Values range from 1-10, and a greater satiety score would be a better outcome in these participants.
Food cravings | Change from baseline to 12 weeks.
  Food cravings as measured by a 10 cm visual analogue scale, where higher values represent greater food cravings. Values range from 1-10, and a greater food cravings score would be a worse outcome in these participants.
Sweet food cravings | Change from baseline to 12 weeks.
  Sweet food cravings as measured by a 10 cm visual analogue scale, where higher values represent greater sweet food cravings. Values range from 1-10, and a greater sweet food cravings score would be a worse outcome in these participants.
Blood urea nitrogen to creatinine ratio | Change from baseline to 12 weeks.
  The ratio of blood urea nitrogen to creatinine in serum.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: No